CLINICAL TRIAL: NCT03636581
Title: A Novel Lifestyle Intervention Program to Improve Body Composition and Chronic Disease Bio Markers in Overweight Medical Students: a Randomized Cross-over Trial
Brief Title: Lifestyle Intervention Program in Overweight Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1333
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive a smart watch to track activity and diet. This group will also receive education on nutrition and exercise.
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention): This group will receive a smart watch to track activity only with no intervention.

INTERVENTIONS:
Behavioral: Lifestyle counseling — This group will receive online education modules to educate them on exercise prescription, nutrition and behavioral changes.
  Arms: Intervention

SUMMARY:
This study will be a randomized cross-over design over the course of 2 academic years. 40 subjects -20 overweight women and 20 over weight men will be recruited. Each subject will have body composition tested, blood lipid profile, and resting metabolic rate done in the beginning of the first academic year and at the end of the first academic year. The intervention group will receive activity trackers, diet counseling, and fitness counseling for one academic year. The second year, all outcome measures (a body scan, blood lipid profile, and resting metabolic rate) will be performed again at the start of the academic year 2, except the intervention group will now be the control group and the control group will now receive the same intervention. All final outcome measures will be performed at the end of the second year.

ELIGIBILITY:
Inclusion Criteria:

* Male and female NYITCOM students between the ages of 18-35
* BMI ≥ 25.0
* Body fat % >19% for males; >33% for women (will be determined by body composition scan)
* Own their own smartphone

Exclusion Criteria:

* People who have used weight loss smartphone applications in the past 6 month
* People who have used an activity tracker in past 6 months
* Anyone who answers yes to one or more questions on the PAR-Q screen
* Any contraindication to having a duel x-ray body scan performed based on the American College of Radiology's practice guidelines

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Body fat percentage | 4 months
  Body composition

SECONDARY OUTCOMES:
Step Count | 4 months
  Activity based on step count
Resting Metabolic Rate | 4 months
  Resting metabolic rate changes as per oxygen consumption
Total Cholesterol | 4 months
  fasting serum mg/dL
High Density Lipoproteins | 4 months
  fasting serum mg/dL
Low Density Lipoproteins | 4 months
  fasting serum mg/dL
Triglycerides | 4 months
  fasting serum mg/dL
Hemoglobin A1C | 4 months
  fasting plasma % of total hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No